CLINICAL TRIAL: NCT03748836
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALPN-101 in Adult Healthy Volunteers
Brief Title: Adult Healthy Volunteers Study to Evaluate ALPN-101 Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AIS-A01
Record Dates: First submitted 2018-11-05; First posted 2018-11-21 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — ALPN-101

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded, dose escalation to evaluate the safety, PK, and PD of single and multiple doses of ALPN-101
Who Masked: Participant, Investigator
Masking Description: Double blinded, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Single Ascending Dose ALPN-101 (Active Comparator)
  Interventions: Drug: ALPN-101
- Single Dose Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Multiple Ascending Dose ALPN-101 (Active Comparator)
  Interventions: Drug: ALPN-101
- Multiple Dose Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALPN-101 — Single or multiple doses of ALPN-101 delivered via intravenous or subcutaneous injection. Ascending dose levels will be evaluated.
  Arms: Multiple Ascending Dose ALPN-101; Single Ascending Dose ALPN-101
Drug: Placebo — Single or multiple doses of placebo delivered via intravenous or subcutaneous injection, matched to ALPN-101 cohorts.
  Arms: Multiple Dose Placebo; Single Dose Placebo

SUMMARY:
This study is testing the safety, tolerability, pharmacokinetics (PK--the amount of study drug in the blood), pharmacodynamics (PD), how the study drug affects the body) and immunogenicity (how the study drug affects the immune system) of single and multiple doses and dose levels of an investigational drug called ALPN-101.

DETAILED DESCRIPTION:
AIS-A01 is a phase 1, randomized, placebo-controlled, double-blinded study in healthy volunteers. It will be conducted at a single center and will enroll approximately 104 participants. The study will have 2 parts:

* In Part A, participants will receive a single dose of study drug or placebo. Multiple dose levels of ALPN-101 will be evaluated.
* In Part B, participants will receive 4 doses of ALPN-101 or placebo--1 dose each week for 4 weeks. Multiple dose levels of ALPN-101 will be evaluated.

In each Part, safety assessments will be performed throughout the dosing and follow-up periods, and multiple PK and PD samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Able to participate and willing to give written informed consent.
2. Healthy adult participant 18 to 65 years of age, inclusive, at the time of informed consent.
3. BMI between 18 and 30 kg/m2, inclusive.
4. Male participants must agree to use a highly effective method of contraception consistently and correctly during the treatment period and for at least 30 days after the last dose of study intervention and to refrain from donating sperm during this period.
5. Female participants must not be pregnant or breastfeeding

   Exclusion Criteria:

   General Health Exclusions
6. Any concomitant disease, condition or treatment that could interfere with the conduct of the study or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the participant in the study or interfere with the interpretation of study data.
7. History or symptoms of significant psychiatric disease in the opinion of the Principal Investigator, including but not limited to depression and schizophrenia.
8. History of immunological disorders, auto-immune disorders, acquired or congenital immune deficiency.
9. History of significant hepatic or renal disease or impairment.
10. Evidence of an active or suspected cancer or a history of malignancy within the previous 3 years, except for the following, which did not require systemic therapy and are considered cured: nonmelanoma skin cancer, curatively treated localised prostate cancer or other in situ cancer.
11. History of major organ transplantation with an existing functional graft. Therapeutic and Intervention-Related Exclusions
12. Use of prescription medications or herbal remedies within 14 days or 5 elimination half-lives (whichever is longer) of study intervention administration or use of over-the-counter medications (OTC) within 7 days of study intervention administration (apart from recommended doses of vitamin/mineral supplements, OTC analgesics, etc., approved by the Investigator and Sponsor). Participants who have been on hormone replacement therapy (HOURST) for a period of at least 2 months will not be excluded from the study, provided the HOURST regimen remains unchanged during the conduct of the study.
13. Any concomitant medications that prolong QT/QTc interval.
14. Dosed with an investigational drug within 30 days or 5 elimination half-lives (whichever is longer) prior to study drug administration.
15. Received any systemic steroid within 1 month or systemic immunosuppressant agent within 6 months prior to study drug administration.
16. Received any antibody therapy or biologic products within 6 months prior to study drug administration.
17. Significant loss of blood including blood donation over 500 mL or transfusion of any blood product within 3 months before the Screening Visit.
18. Unwilling to refrain alcohol use 48 hours prior to your admission into the clinical research unit.
19. Known hypersensitivity, allergy or intolerance to the study drug or any of the excipient contained in the intervention formulation.
20. Immunisation with any vaccine within 6 weeks prior to study drug administration.
21. For participants enrolled in cohorts in which KLH will be administered: known administration of KLH within 6 months prior to study drug administration; known seafood or shellfish allergy, or known hypersensitivity or allergy to KLH Laboratory Exclusions
22. Any clinically significant (at the discretion of the Investigator) abnormalities in laboratory test results, including complete blood count, chemistry panels and urinalysis. If out of range at the Screening Visit and/or admission to the CRU and deemed clinically significant by investigator, the tests may be repeated once on a separate day.
23. Estimated creatinine CL < 90 mL/minute at the Screening Visit
24. Positive test at the Screening Visit and/or at baseline for drugs of abuse (e.g., phencyclidine, opiates, benzodiazepines, barbiturates, amphetamines, methamphetamines, cocaine and THC). The repeat test is permitted once for a suspected false positive test.
25. Positive alcohol breath test at the Screening Visit and/or at baseline.
26. Positive result on tests for HIV-1 and/or HIV-2 antibody, anti-hepatitis B virus antibodies (core antibody [HBcAb], surface antigen [HBsAg]) or anti-hepatitis C virus antibody.
27. Positive serum pregnancy test at the Screening Visit or admission to the CRU. Infection-related Exclusions.
28. Acute infection including viral infections in the preceding 6 weeks
29. History or presence of any chronic infectious condition, including but not limited to tuberculosis or parasitic infections. Evidence of tuberculosis may include either a positive tuberculosis blood test (by a positive QuantiFERON® TB-Gold test or a positive tuberculin skin test) or chest X-ray radiographic findings consistent with active or latent tuberculosis.

    Cardiovascular Exclusions
30. Supine sustained (i.e. 3 independent measurements within 30 min) systolic blood pressure greater than 140 or less than 90 mmHg.
31. Supine sustained (i.e. 3 independent measurements within 30 min) diastolic blood pressure greater than 90 or less than 40 mmHg.
32. Sustained (i.e. 3 independent measurements within 30 min) heart rate (pulse) greater than 100 or less than 40 beats per minute (bpm).
33. QTcF < 300 msec or ≥ 450 msec.
34. Personal and/or family history of congenital long QT syndrome or sudden cardiac death

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Safety, as assessed by adverse events according to CTCAE v5.0 | From study Day 1 (dosing of ALPN-101 or placebo) until the End of Study visit (approx. 4-8 weeks)
  The rate of adverse events will be compared between the 2 treatment groups.

SECONDARY OUTCOMES:
Pharmacokinetics of ALPN-101 as assessed by time of maximum ALPN-101 concentration. | From study Day 1 (dosing of ALPN-101 or placebo) until the End of Study visit (approx. 4 weeks for Part A of the study, and approx 6 weeks for Part B)
  Plasma levels of ALPN-101 will be serially evaluated following dosing of study drug, and the time of maximum plasma concentration (Tmax) will be identified.
Pharmacokinetics of ALPN-101 as assessed by the maximum concentration of ALPN-101. | From study Day 1 (dosing of ALPN-101 or placebo) until the End of Study visit (approx. 4 weeks for Part A of the study, and approx 6 weeks for Part B)
  Plasma levels of ALPN-101 will be serially evaluated following dosing of study drug, and the maximum plasma concentration (Cmax) will be calculated.
Pharmacokinetics of ALPN-101 as assessed by AUC on all subjects. | From study Day 1 (dosing of ALPN-101 or placebo) until the End of Study visit (approx. 4 weeks for Part A of the study, and approx 6 weeks for Part B)
  Plasma levels of ALPN-101 will be serially evaluated following dosing of study drug, and the area under the curve (AUC) will be calculated.
The incidence of ADA against ALPN-101 will be assessed and summarized. | From study Day 1 (dosing of ALPN-101 or placebo) until the End of Study visit (approx. 4 weeks for Part A of the study, and approx 6 weeks for Part B)
  The incidence of ADA against ALPN-101 will be assessed by the percentage of patients with a positive ADA result of all the treated patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network- Centre for Clinical Studies, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No